CLINICAL TRIAL: NCT00764244
Title: VITRILASE Study: Prospective Randomized Trial Comparing the Effect of Laser, Vitrectomy and Intravitreal Triamcinolone Injection for Diabetic Macular Edema
Brief Title: Laser Versus Vitrectomy Versus Intravitreal Triamcinolone Injection for Diabetic Macular Edema
Acronym: VITRILASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P030426; MUL03010
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2014-11

CONDITIONS: Diabetic Macular Edema; Diabetes
Keywords: Diabetes; Macular edema; Optical Coherence tomography; VitrectomyLaser therapy; Intravitreal triamcinolone injection
MeSH Terms: conditions — Diabetes Mellitus; Macular Edema | interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Vitrectomy
  Interventions: Procedure: Vitrectomy
- 2 (Active Comparator): Intravitreal triamcinolone injections
  Interventions: Drug: Intravitreal triamcinolone injections
- 3 (Active Comparator): Laser photocoagulation
  Interventions: Procedure: Laser photocoagulation

INTERVENTIONS:
Procedure: Vitrectomy — Vitrectomy
  Arms: 1
Drug: Intravitreal triamcinolone injections — Intravitreal triamcinolone injections
  Other Names: - KENACORT RETARD; - Triamcinolone Acetonid
  Arms: 2
Procedure: Laser photocoagulation — Laser photocoagulation
  Arms: 3

SUMMARY:
Macular edema is the main cause of vision loss in diabetic patients. Its treatment is mainly based on laser photocoagulation, but has limited results. Alternative treatment are under investigation, such as vitrectomy and intravitreal injections of triamcinolone .The aim of VITRILASE is to compare the efficacy of these two treatments to laser photocoagulation for diabetic macular edema.

DETAILED DESCRIPTION:
It is a randomized study with three arms

* vitrectomy
* repeat intravitreal triamcinolone injections
* laser photocoagulation

ELIGIBILITY:
Inclusion Criteria:

1. Patient with type 1 or type 2 diabetes
2. Visual acuity (VA) : 0.1≤ VA < 0.5 (35 ≤ ETDRS score < 70)
3. Patient with diffuse diabetic macular edema , as defined by :§ Retinal thickening involving the center of the macular on biomicroscopy§ AND diffuse leakage on fluorescein angiography .
4. Macular thickness in the central area 1000 µm in diameter ³ 300 µm.
5. Patient with :· Either diffuse diabetic macular edema · Or combined diffuse and focal diabetic macular edema with persistent diffuse macular edema 6 months after laser treatment of the focal edema .
6. Systolic blood pressure ≤ 160 mmHg and diastolic blood pressure ≤ 90 mmHg.,
7. HbA1c < 10%.

Exclusion Criteria:

1. Patient with tractional diabetic macular edema, as defined by· A taut, thickened posterior hyaloid on biomicroscopy AND/OR· a thickened , highly reflective posterior hyaloid on OCT , partially detached from the posterior pole, and exerting a traction on the macula
2. Active proliferative diabetic retinopathy (ETDRS stage 61 or more severe)
3. Structural damage to the center of the macula in the study eye likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s), or organized central hard exudate plaque³ 1 disk area
4. Hypertensive retinopathy
5. Epiretinal membrane.
6. Rubeosis irides .
7. Patient requiring immediate panretinal photocoagulation or panretinal photocoagulation performed within the past 6 months .
8. History of chronic glaucoma in the study eye
9. History of elevated intraocular pressure ≥30 mm Hg and/or alteration of visual field
10. Concomitant therapy with systemic or topical ocular corticosteroids within the last 15 days .
11. Cataract surgery in the study eye within the past 6 months, Yttrium-Aluminum-Garnet (YAG) laser capsulotomy within the past 6 months,
12. Aphakia
13. Patient with pseudophakic macula edema
14. Unstable medical status including glycemic control and blood pressure. Patients in poor glycemic control who, within the last 4 months, initiated intensive insulin treatment (a pump or multiple daily injections) should not be enrolled.
15. Chronic renal failure
16. Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2005-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with visual gain ≥ 3 ETDRS lines at 2 years | at 2 years

SECONDARY OUTCOMES:
Central macular thickness on Optical Coherence Tomography (OCT) | at 8, 12 and 24 months
Percentage of patients with visual gain ≥ 3 ETDRS lines | 8, 12 and 22 months
Progression of lens opacities | During the all follow-up
Frequency of complications | During the all follow-up
Results analysis according to preoperative vitreous detachment, honeycomb macular edema on fluorescein angiography | at inclusion time
Evolution of visual fiends and posterior vitreous detachment | At inclusion time and 2 years
Percentage of patients presenting an increase of 2 line or more of best corrected visual acuity on ETDRS charts | after 1 year, 22 months and 24 months of follow-up
Percentage of patients presenting an decrease of 2 line or more of best corrected visual acuity on ETDRS charts | after 1 year, 22 months and 24 months of follow-up
Scores ETDRS | after 1 year, 22 months and 24 months of follow-up
Mean best corrected visual acuity during follow-up period | during the all follow-up
Progression of retinopathy diabetic in each group | during the all follow-up
Outcome in respect to posterior vitreal detachment (PVD) stage | during the all follow-up
PVD stage evolution during the follow-yp in laser and triamcinolone group | first and last exam
Evolution of visual field in each group | inclusion and last visit

CONTACTS AND LOCATIONS:
Overall Officials: Pascale MASSIN, MD, PhD; Pr, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Pascale MASSIN, Paris, France

REFERENCES:
- [Result] Audren F, Lecleire-Collet A, Erginay A, Haouchine B, Benosman R, Bergmann JF, Gaudric A, Massin P. Intravitreal triamcinolone acetonide for diffuse diabetic macular edema: phase 2 trial comparing 4 mg vs 2 mg. Am J Ophthalmol. 2006 Nov;142(5):794-99. doi: 10.1016/j.ajo.2006.06.011. Epub 2006 Sep 15. PMID 16978576